CLINICAL TRIAL: NCT05114720
Title: A Multicenter, Placebo-Controlled, Phase III Trial of Standard Adjuvant Chemotherapy Plus Moxifloxacin in Operable Breast Cancer
Brief Title: Moxifloxacin in Adjuvant Treatment of Patients With Operable Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Professor of Medicine, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSUCC-015
Record Dates: First submitted 2021-11-02; First posted 2021-11-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: moxifloxacin; operable breast cancer; adjuvant treatment; disease-free survival; safety
MeSH Terms: conditions — Breast Neoplasms | interventions — Moxifloxacin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard adjuvant chemotherapy plus moxifloxacin (Experimental): Standard adjuvant chemotherapy (Taxanes combined with cyclophosphamide or doxorubicin combined with cyclophosphamide followed by taxanes) plus antibiotic (moxifloxacin)
  Other Name: docetaxel 75mg/m^2, or nab-paclitaxel 260mg/m^2, IV, days 1, cycled every 21 days cyclophosphamide 1000 mg/m^2, IV, days 1, cycled every 21 days; or doxorubicin 60mg/m^2, IV, days 1, combined with cyclophosphamide 600 mg/m^2, IV, days 1, followed by docetaxel 75mg/m^2, or nab-paclitaxel 260mg/m^2, IV, days 1; plus Moxifloxacin 0.4 PO once daily days 1-5; cycled every 21 days
  Interventions: Drug: standard adjuvant chemotherapy plus moxifloxacin
- standard adjuvant chemotherapy plus placebo (Placebo Comparator): Standard adjuvant chemotherapy (Docetaxel combined with cyclophosphamide or doxorubicin combined with cyclophosphamide followed by docetaxel) plus placebo
  Other Name: docetaxel 75mg/m^2, or nab-paclitaxel 260mg/m^2, IV, days 1 cyclophosphamide 1000 mg/m^2, IV, days 1, cycled every 21 days; or doxorubicin 60mg/m^2, IV, days 1, combined with cyclophosphamide 600 mg/m^2, IV, days 1, followed by docetaxel 75mg/m^2, or nab-paclitaxel 260mg/m^2, IV, days 1; plus Placebo 0.4 PO once daily days 1-5; cycled every 21 days
  Interventions: Drug: standard adjuvant chemotherapy plus placebo

INTERVENTIONS:
Drug: standard adjuvant chemotherapy plus moxifloxacin — docetaxel 75mg/m^2, or nab-paclitaxel 260mg/m^2, IV, days 1 cyclophosphamide 1000 mg/m^2, IV, days 1, cycled every 21 days; or doxorubicin 60mg/m^2, IV, days 1, cycled every 21 days cyclophosphamide 600 mg/m^2, IV, days 1, cycled every 21 days docetaxel 100 mg/m^2, IV, days 1, cycled every 21 days; plus Moxifloxacin 0.4 PO once daily days 1-5; cycled every 21 days
  Other Names: Standard adjuvant chemotherapy (Docetaxel combined with cyclophosphamide or doxorubicin combined with cyclophosphamide followed by docetaxel) plus antibiotic (moxifloxacin)
  Arms: standard adjuvant chemotherapy plus moxifloxacin
Drug: standard adjuvant chemotherapy plus placebo — docetaxel 75mg/m^2, or nab-paclitaxel 260mg/m^2, IV, days 1 cyclophosphamide 1000 mg/m^2, IV, days 1, cycled every 21 days; or doxorubicin 60mg/m^2, IV, days 1, cycled every 21 days cyclophosphamide 600 mg/m^2, IV, days 1, cycled every 21 days docetaxel 100 mg/m^2, IV, days 1, cycled every 21 days; plus Placebo 0.4 PO once daily days 1-5; cycled every 21 days
  Other Names: Standard adjuvant chemotherapy (Docetaxel combined with cyclophosphamide or doxorubicin combined with cyclophosphamide followed by docetaxel) plus placebo
  Arms: standard adjuvant chemotherapy plus placebo

SUMMARY:
The primary objective of this study is to compare disease-free survival (DFS) of patients with operable breast cancer randomised to treatment with standard adjuvant chemotherapy plus moxifloxacin or placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomised, double-blind, placebo-controlled, phase 3 clinical trial. The main purposes of this study are to examine the efficacy and safety of standard adjuvant chemotherapy plus moxifloxacin or placebo as care for patients with operable breast cancer. This study is designed to recruit up to 520 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written and signed informed consent;
2. Histologically confirmed invasive ductal carcinoma;
3. Planned to received (neo)/adjuvant chemotherapy;
4. Eastern Cooperative Oncology Group (ECOG) score of 0 to 1;
5. Normal blood routine, liver and kidney functions within 1 week before enrollment in this study;
6. Women of childbearing age have a negative serum or urinary pregnancy tests prior to enrollment in this study; Pre-menopause women are contracepted with medically acceptable methods during the study period.
7. Compliance with the study protocol.

Exclusion Criteria:

1. Pregnant or breast feeding;
2. Eastern Cooperative Oncology Group (ECOG) score ≥ 2;
3. Hypersensitivity to moxifloxacin or quinolones compounds;
4. Concomitant with other antitumor therapies or participating in other clinical trials;
5. Have a history of heart disease, such as arrhythmia, conduction block, S-T segment elevation, ischemic heart disease, or congenital heart disease;
6. Severe uncontrolled co-infection, or severe metabolic disorders;
7. A clear past history of neurological or psychiatric disorders, including epilepsy or dementia;
8. Poor compliance, unwillingness or inability to follow protocol to continue the study;
9. Any circumstances in which the investigator deemed the subject unsuitable for enrollment in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 10 years
  The interval from the date of randomization until the first date of recurrence local, regional or distant, second primary tumor or death due to any cause

SECONDARY OUTCOMES:
overall survival (OS) | 10 years
  The interval from the date of randomization until the first date on death due to any cause, or the last follow-up time
distant disease-free survival (DDFS) | 10 years
  The interval from the date of randomization until the first date on distant metastasis, death due to any cause, or second primary invasive breast cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
We decided to not share our individual participant data (IPD) to other researchers.